CLINICAL TRIAL: NCT03354182
Title: Treatment of Mandibular Type II Furcations Using Bovine-derived Bone Xenograft With or Without a Collagen Membrane: a Randomized Clinical Trial
Brief Title: Surgical Treatment of Mandibular Furcations Using a Xenograft With/Without a Collagen Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/03AVR/167
Record Dates: First submitted 2017-10-19; First posted 2017-11-27 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-06

CONDITIONS: Furcation Defects
Keywords: Mandibular type II furcations; Periodontal treatment; Demineralized bovine bone mineral; Collagen membrane
MeSH Terms: conditions — Furcation Defects

STUDY DESIGN:
Intervention Model Description: Randomized clinical study with 1 control group and 1 test group
Who Masked: Participant
Masking Description: The patients didn't know whether they were the control or test group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Open flap surgery on mandibular type II furcations treated with Bio-oss collagen + Bio-gide
  Interventions: Procedure: Open flap surgery; Device: Bio-oss collagen; Device: Bio-gide
- Test group (Active Comparator): Open flap surgery on mandibular type II furcations treated with Bio-oss collagen alone
  Interventions: Procedure: Open flap surgery; Device: Bio-gide

INTERVENTIONS:
Procedure: Open flap surgery — Elevation of a flap in order to access the treated furcation
Device: Bio-oss collagen — Biomaterial for periodontal surgery
  Arms: Control group
Device: Bio-gide — Biomaterial for periodontal surgery

SUMMARY:
The aim of the study was to perform a randomized controlled clinical study in order to compare the effects of a bovine derived xenograft (with 10% collagen) + a bioabsorbable membrane (control group, CG) vs a bovine derived xenograft (with 10% collagen) alone (test group, TG) on the surgical treatment of mandibular type II furcation defects.

DETAILED DESCRIPTION:
The aim of the study was to perform a randomized controlled clinical study in order to compare the effects of a bovine derived xenograft (with 10% collagen) + a bioabsorbable membrane (control group, CG) vs a bovine derived xenograft (with 10% collagen) alone (test group, TG) on the surgical treatment of mandibular type II furcation defects. The patients all underwent the same surgical intervention with the only difference between the two groups being the use or not of a collagen membrane.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic periodontitis
* Initial phase (oral hygiene instructions + full mouth scaling and root planing) performed at least eight weeks before inclusion
* Full-mouth plaque score ≦ 20% (at least eight weeks after initial phase and during the whole treatment)
* Clinical evidence of vestibular or lingual mandibular Class II furcation defects (≧ 3mm of horizontal probing depth)
* Presence of at least 2 mm of keratinized gingiva on the selected tooth surface facing the furcation
* Tooth vitality confirmed by clinical tests (cold testing)

Exclusion Criteria:

* Presence of any systemic disease
* Smokers
* Devitalized tooth or tooth presenting periapical or pulpar pathology (confirmed with a retro-alveolar radiograph)
* Allergies to any of the products used in the present study
* Pregnant or breastfeeding women
* History or current RX therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-07-30 (Actual); Primary Completion 2017-01-02 (Actual); Study Completion 2017-01-02 (Actual)

PRIMARY OUTCOMES:
Horizontal Probing Attachment Level | 6 months
  PAL-H